CLINICAL TRIAL: NCT06072417
Title: Comparative Study of Sleep Disordered Breathing (SDB) in Patients With Pulmonary Vascular Diseases Permanently Residing Above 2500 Meters When Assessed Near Resident High Altitude (HA) at 2840m vs. at Low Altitude (LA) Sea Level
Brief Title: HA Residents With PVD, SDB Assessed at HA (2840m) vs LA (Sea Level)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PVD_HAvsLA_SDB
Record Dates: First submitted 2023-08-09; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Vascular Disease; Pulmonary Artery Hypertension; Chronic Thromboembolic Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Hypoxia; sleep disordered breathing; Pulmonary arterial hypertension; Chronic Thromboembolic Pulmonary Hypertension; High altitude
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Hypertension, Pulmonary; Hypoxia; Sleep Apnea Syndromes; Pulmonary Arterial Hypertension; Altitude Sickness | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Patients living permanently >2500m around Quito (Equador) will be assessed at 2840m and after relocation to sea level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory sleep study at 2840m (Placebo Comparator): Participants will have a respiratory sleep study by polygraphy near their resident altitude at 2840m
  Interventions: Other: Assessment without intervention at High altitude
- Respiratory sleep study near sea level (0-30m) (Experimental): Participants will have a respiratory sleep study by polygraphy near sea level (0-30m)
  Interventions: Other: Relocation to sea level for 2 days

INTERVENTIONS:
Other: Assessment without intervention at High altitude — Assessments at High altitude corresponding to Baseline measures
  Arms: Respiratory sleep study at 2840m
Other: Relocation to sea level for 2 days — Participants will be relocated to sea level and intervention and have assessements there.
  Arms: Respiratory sleep study near sea level (0-30m)

SUMMARY:
To study the effect of relocation from 2840m (Quito) to sea level (Pedernales) in patients with pulmonary vascular diseases (PVD) defined as pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension (PH) who permanently live >2500m on sleep disordered breathing

DETAILED DESCRIPTION:
This research in patients with PVD diagnosed with precapillary PH with right heart catheterization and classified to groups 1 and 4 (PAH or CTEPH) who permanently live at HA >2500 (PVDHA) will have nocturnal respiratory sleep studies near their living altitude in Quito at 2840m and at sea level in Pedernales during the first and the second night after relocation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-80 years old of both genders,
* Residence > 2500m of altitude
* diagnosed with precapillary PH (mean pulmonary artery pressure (mPAP) >20 mmHg, pulmonary artery wedge pressure (PAWP) ≤15 mmHg and pulmonary vascular resistance (PVR) ≥2 WU (wood units) by right heart catheterization) with PH being classified as PAH or CTEPH according to guidelines
* Patients stable on therapy
* NYHA (new york heart association) functional class I-III
* Provided written informed consent to participate in the study.

Exclusion Criteria:

* Age <18 years or >80 years
* unstable condition
* Patients who cannot follow the study investigations, patient permanently living < 2500m.
* Patients with moderate to severe concomitant lung disease (FEV1<70% or forced vital capacity <70%), severe parenchymal lung disease, severe smokers (>20 cigarettes/day)
* Severely hypoxemic patients at Quito permanently have persistent SpO2 (oxygen saturation by pulseoximetry) <80% on ambient air.
* Patients with chronic mountain sickness (Hemoglobin > 19 g/dl in women, >21 g/dl in men)
* Patient with a non-corrected ventricular septum defect
* Relevant concomitant other disease of the heart, kidney, liver, blood (anemia hemoglobin<11 g/dl)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean nocturnal SpO2 at LA vs. HA | during the first night at low altitude (of intervention)
  Change in mean nocturnal SpO2 (%) between LA (sea level) vs HA (2840 m)

SECONDARY OUTCOMES:
Mean nocturnal SpO2 at LA vs. HA | during the second night at low altitude (of intervention)
  Change in mean nocturnal SpO2 (%) between LA (sea level) vs HA (2840 m)
Time spent with SpO2<90% at LA vs. HA | during the first and second night at low altitude (of intervention)
  Change in time spent with SpO2<90% between LA (sea level) vs HA (2840 m)
AHI at LA vs. HA | during the first and second night at low altitude (of intervention)
  Change in apnea-hypopnea index (AHI) between LA (sea level) vs HA (2840 m)
ODI at LA vs. HA | during the first and second night at low altitude (of intervention)
  Change in oxygen desaturation index (ODI) between LA (sea level) vs HA (2840 m)
Time spent with periodic breathing at LA vs. HA | during the first and second night at low altitude (of intervention)
  Change in time spent with periodic breathingbetween LA (sea level) vs HA (2840 m)
Heart rate variability at LA vs. HA | during the first and second night at low altitude (of intervention)
  Change in heart rate variability between LA (sea level) vs HA (2840 m)
ECG markers of repolarization at LA vs. HA | during the first and second night at low altitude
  Change in electrocardiogram (ECG) markers of repolarization (QT time) between LA (sea level) vs HA (2840 m)
pulse transit time drops at LA vs. HA | during the first and second night at low altitude
  Change in pulse transit time drops between LA (sea level) vs HA (2840 m)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, Prof. Dr., Principal Investigator — University Hospital Zurich, Departement of Pulmonology; Rodrigo Hoyos, Dr., Principal Investigator — Carlos Adrade Marin Hospital of Quito, Equador
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data will be provided upon request and based on a clear intention reviewed by an ethical review board.